CLINICAL TRIAL: NCT04366531
Title: Development of a Psycho-social Transition Program and Transition Assessment Tools for Veterans With Mental Illness and/or Substance Use Disorders Leaving Prison
Brief Title: Successful Transitions and Reintegration Tools for Veterans (START-VETS)
Acronym: START-VET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3225-R
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Substance Use Disorder; Mental Illness; Recently Incarcerated
Keywords: reentry; Mental illness; prison; substance use disorder
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Veterans will be randomly assigned to either begin an eight week (actual number of weeks is to be determined based on phase 2) active treatment program or to a no treatment phase. At eight weeks veterans will switch the condition they were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monitoring/Treatment as usual (No Intervention): Veterans will not receive any study related interventions.
- Reentry Program (Active Comparator): Veterans will receive the START-VET reentry program
  Interventions: Behavioral: START-VET; Other: Treatment as usual

INTERVENTIONS:
Behavioral: START-VET — prison reentry program
  Arms: Reentry Program
Other: Treatment as usual — This intervention involves no additional services above what is provided by the local health care system
  Arms: Reentry Program

SUMMARY:
This study will develop prison reentry materials for Veterans leaving prison.

DETAILED DESCRIPTION:
This study will be conducted in three phases Phase 1 is to collect qualitative data from Veterans who have recently been released from prison. The data will focus on their transition experience, stigma (both self and from others), and behaviors that interfered with success.

Phase 2a will be to develop a transition program based around the needs identified in phase 1 Phase 2b will be to develop assessment tools to be used with the program Phase 3 will be to perform a two group randomized cross over design pilot study to assess the program

ELIGIBILITY:
Inclusion Criteria:

* Veteran with mental illness and/or substance use disorder released from prison within the past 36 months

Exclusion Criteria:

* psychosis or cognitive impairment precluding active participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Brief Symptom Inventory -18 | The Brief Symptom Inventory will be administered at the baseline of the subject's participation and again every 4 weeks for 16 weeks.
  The Brief Symptom Inventory - 18 evaluates the domains of Somatization, Depression, and Anxiety. Each scale has 6 items, with a range of 0-24. Higher indicates a higher amount of the identified construct, i.e a worse outcome.
Change in the World Health Organization Quality of Life 100 | The World Health Organization Quality of Live 100 will be administered at the baseline of the subject's participation and again every 4 weeks for 16 weeks.
  The World Health Organization Quality of Life 100 is a overall measure quality of life for participants. It has 5 domains: Physical (12 items, range 12-60), Psychological (18 items, range 18-90), Independence (16 items, range 16 - 80), Social (12 items, range 12-60), Environment (32 items, range 32-160), and Spiritual (4 items, range 4-20). Higher indicates higher levels of quality of life.
Inventory of Criminal Thinking Style | The Inventory of Criminal Thinking Style will be administered at the baseline of the subject's participation and again every 4 weeks for 16 weeks.
  The Inventory of Criminal Thinking Styles (PICTS) is an 80-item self-report inventory designed to measure eight thinking styles presumed to reinforce, support, and maintain a criminal lifestyle. The eight thinking styles assessed by the PICTS are Mollification, Cutoff, Entitlement, Power Orientation, Superoptimism, Sentimentality, Cognitive Indolence, and Discontinuity. There are 10 items on each scale with scale scores ranging from 0 - 30. Higher indicates worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: James P. LePage, PhD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (1):
- VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No